CLINICAL TRIAL: NCT07032051
Title: Preventive Effects of Continuous Passive Motion on Ankle Contracture and Muscle Atrophy in Mechanically Ventilated Patients: A Pilot Study
Brief Title: Continuous Passive Motion to Prevent Ankle Contracture and Muscle Atrophy in Ventilated Patients
Acronym: CPM-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPM-SKH-20240808R; 20240808R (Other: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Ankle Contracture; Critically Ill Intensive Care Unit Patients; Muscle Atrophy
Keywords: ICU-acquired weakness; muscle ultrasound; ankle contracture; continuous passive motion,
MeSH Terms: conditions — Muscular Atrophy | interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Intervention Model Description: This study uses a within-subject controlled design with a single-group assignment model. Each participant receives continuous passive motion (CPM) therapy on the left ankle, while the right ankle, without CPM, serves as the control. This approach enables direct comparison of outcomes between the intervention and control conditions within the same individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPM Intervention Group (Experimental): All participants received continuous passive motion (CPM) therapy on the left ankle once daily for seven consecutive days during mechanical ventilation. The right ankle, which did not receive CPM, served as the within-subject control. This single-arm trial employed a within-subject controlled design to allow direct comparison between the treated and untreated limbs in the same individual.
  Interventions: Device: Continuous Passive Motion

INTERVENTIONS:
Device: Continuous Passive Motion — Continuous passive motion was applied to the left ankle joint for 30 minutes twice a day using a motorized CPM device.

SUMMARY:
This clinical trial aims to evaluate whether continuous passive motion (CPM) can prevent ankle joint contracture and muscle atrophy in critically ill patients receiving mechanical ventilation in the ICU. The study will also assess the feasibility and safety of implementing CPM therapy in this population.

The primary objectives are:

To determine whether CPM preserves ankle dorsiflexion range of motion during ICU immobilization.

To assess whether ultrasound can detect changes in tibialis anterior muscle morphology in response to CPM.

In this within-subject design, each participant will receive CPM therapy on one ankle while the contralateral ankle serves as the control. Outcomes related to joint mobility and muscle condition will be compared between the two sides.

Participants will:

Receive CPM treatment on one ankle for 30 minutes, twice daily, for up to 7 days or until ICU discharge.

Undergo goniometric and ultrasound assessments at baseline and after the intervention.

Continue to receive standard ICU care throughout the study period.

DETAILED DESCRIPTION:
Critically ill patients commonly experience neuromuscular complications, notably intensive care unit-acquired weakness (ICU-AW) and joint contractures. ICU-AW affects up to 80% of patients requiring prolonged mechanical ventilation and is associated with prolonged hospitalization, delayed functional recovery, and increased mortality. Concurrently, immobility during ICU stays contributes significantly to joint contractures, affecting approximately one-third of patients experiencing extended ICU admissions. Among these complications, ankle joint plantar-flexion contractures (foot drop) are particularly debilitating, severely impacting patients' balance, gait retraining, and overall functional recovery after ICU discharge.

Although early mobilization is widely recognized as beneficial, leading to reduced ICU stays, lower incidence of delirium, preservation of muscle integrity, and enhanced quality of life post-discharge, its implementation remains challenging. Many critically ill patients are unable to participate in early active mobilization due to sedation, hemodynamic instability, or other medical contraindications. Furthermore, evidence suggests that early mobilization might carry increased risks of adverse events for certain patient populations. Thus, alternative strategies are essential for patients unsuitable for early active rehabilitation, emphasizing preservation of joint mobility and muscle integrity to facilitate future rehabilitation opportunities.

Continuous passive motion (CPM) therapy has emerged as a viable intervention designed initially for postoperative orthopedic rehabilitation. CPM passively moves joints through a controlled range, potentially maintaining flexibility by inhibiting periarticular collagen cross-linking, preserving soft tissue extensibility, and maintaining muscle-tendon compliance. However, its effectiveness in critical illness settings remains uncertain, with limited evidence suggesting potential benefits in reducing muscle atrophy, such as that of the tibialis anterior muscle, in ICU patients unable to actively mobilize, while other studies have reported minimal effects. Thus, rigorous evaluation of CPM's impact on joint mobility preservation and muscle atrophy prevention is warranted.

This study aimed to evaluate whether CPM therapy effectively mitigates passive range of motion (PROM) loss at the ankle joint in sedated, mechanically ventilated ICU patients. Additionally, muscle structural changes were assessed via ultrasound imaging to determine if CPM influences muscle morphology compared to limbs receiving standard care alone. Ultrasound parameters, including muscle thickness (MT), cross-sectional area (CSA), echointensity (EI), and pennation angle (PA), were used to comprehensively monitor morphological changes and provide insights into the functional implications of observed alterations.

ELIGIBILITY:
Inclusion Criteria:

- Eligible participants were adults (≥18 years) with acute respiratory failure expected to require mechanical ventilation for >5 days.

Exclusion Criteria:

* Neuromuscular disorders
* Recent lower limb surgery or trauma
* Critical limb ischemia
* Limb amputation
* Deep vein thrombosis
* Significant leg wounds
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Passive Ankle Dorsiflexion Range of Motion (ROM) | Baseline and Day 7 or until ICU discharge
  Difference in passive ankle dorsiflexion angle between baseline and Day 7, measured using a goniometer. The left (intervention) and right (control) ankles will be compared within each subject. Reported in degrees (°).

SECONDARY OUTCOMES:
Tibialis Anterior Muscle Thickness | Baseline and Day 7
  Change in muscle thickness of the tibialis anterior as measured by ultrasound. Measurements will be obtained directly from B-mode ultrasound images using the built-in caliper function of the ultrasound machine. Values will be reported in centimeters (cm).
Tibialis Anterior Muscle Cross-section Area | Baseline and Day 7
  Change in cross-sectional area of the tibialis anterior muscle as measured by ultrasound. Measurements will be obtained directly using the built-in area tracing tool on the ultrasound machine during B-mode imaging. Values will be reported in square centimeters (cm²).
Tibialis Anterior Muscle Echointensity | Baseline and Day 7
  Change in echointensity of the tibialis anterior muscle as measured from B-mode ultrasound images. Echointensity will be quantified using ImageJ software as the mean and standard deviation of grayscale values within a manually selected region of interest (ROI), ranging from 0 (black) to 255 (white). Reported in grayscale arbitrary units (AU).

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-su Memorial Hospital, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No